CLINICAL TRIAL: NCT04404855
Title: Randomized Clinical Trial Using Next Generation Microbial Sequencing to Direct Antibiotic Selection Before Kidney Stone Lithotripsy Using an Interprofessional Model
Brief Title: Antibiotic Selection Using Next Generation Sequencing vs Urine Culture
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Microgen LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC20190678H
Record Dates: First submitted 2020-05-13; First posted 2020-05-28 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Kidney Stone; Renal Stone; Infection, Bacterial
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Parallel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (NGS + Antibiotic Recommendation) (Other): Next Generation Sequencing results along with Infectious Disease Pharmacist will be shared with clinical provider to determine appropriate standard of care antibiotic treatment at time of standard of care urology stone procedure. Standard of care antibiotic selection will be up to the discretion of the clinical provider.
  Interventions: Other: NGS + Antibiotic Recommendation
- Control Group (Other): NGS results will not be shared with the clinical provider at time of standard of care urology stone procedure. Standard of care antibiotic selection will be up to the discretion of the clinical provider.
  Interventions: Procedure: Standard of Care treatment

INTERVENTIONS:
Other: NGS + Antibiotic Recommendation — NGS results in addition to recommended antibiotic therapy made by infectious disease pharmacist
  Arms: Intervention Group (NGS + Antibiotic Recommendation)
Procedure: Standard of Care treatment — Subjects will have a standard of care urine culture and prophylactic antibiotic prescribed per routine care.
  Arms: Control Group

SUMMARY:
This is a randomized controlled clinical study evaluating the use of next-generation sequencing (NGS) to improve antibiotic prescribing before ureteroscopy or percutaneous nephrolithotomy.

DETAILED DESCRIPTION:
NGS will be performed on voided urine collected as routine care approximately 30 days prior to surgery. Results will be presented to Infectious Disease pharmacist within 48-72 hours to help select the most appropriate antibiotics, and independently as part of routine care, surgeons will choose the antibiotic that they would use in each case, while the Infectious Disease pharmacists would select their optimum choice. Approximately 220 subjects will be randomly assigned in a 1:1 ratio to receive either NGS antibiotic recommendation or standard of care (SOC) prophylaxis prescribed treatment. Subjects assigned to standard of care will have urine cultures sent for analysis, and the physician will choose antibiotics based on results as per usual practice. Subjects assigned to the NGS group, in addition to routine urine culture results, will have NGS urine culture results sent to an investigational drrug (ID) pharmacist, and recommendations will be shared with the physician to determine the antibiotic selection. The physician will ultimately decide the appropriate antibiotics to prescribe. Approximately 7-14 days after surgery, the research staff will conduct a telephone call to ask about any post-operative infections, complications, and any additional antibiotics that were prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Patients planning to undergo kidney or bladder stone removal surgery using endoscopy including ureteroscopy and percutaneous nephrolithotomy or any other transurethral procedure
* Age 18 or older
* Able to give informed consent

Exclusion Criteria:

* Unwilling or unable to provide informed consent
* Age < 18
* Does not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Liss, MD, Principal Investigator — University of Texas Health at San Antonio
Locations (3):
- United States (3):
  - Audie Murphy VA Hospital, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, Medical Arts and Research Center, San Antonio, Texas
  - University Health System, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data be shared, in addition to the individual participant data set and data dictionaries for the IPD itself.
Supporting Information: Study Protocol, SAP
Time Frame: At the time of publication in a peer review journal

REFERENCES:
- [Result] Liss MA, Reveles KR, Tipton CD, Gelfond J, Tseng T. Comparative Effectiveness Randomized Clinical Trial Using Next-generation Microbial Sequencing to Direct Prophylactic Antibiotic Choice Before Urologic Stone Lithotripsy Using an Interprofessional Model. Eur Urol Open Sci. 2023 Sep 28;57:74-83. doi: 10.1016/j.euros.2023.09.008. eCollection 2023 Nov. PMID 38020524
- See also: Comparative Effectiveness Randomized Clinical Trial Using Next-generation Microbial Sequencing to Direct Prophylactic Antibiotic Choice Before Urologic Stone Lithotripsy Using an Interprofessional Model — https://doi.org/10.1016/j.euros.2023.09.008

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Group (NGS + Antibiotic Recommendation) | Control Group
Started | 119 | 121
Completed | 50 | 86
Not Completed | 69 | 35
Not completed — Subjects who did not complete were either screened positive for infection or non compliant | 69 | 35

BASELINE CHARACTERISTICS:
Population: 50 subjects from the intervention group were included in the analysis population and 86 in the control group. Other subjects were screen failures or non-compliant with study procedures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group (NGS + Antibiotic Recommendation) | Control Group | Total
Number analyzed (Participants) | 50 | 86 | 136
Age, Continuous [Median (Full Range); unit: years] | 50 [40 to 61] | 52 [41 to 66] | 52 [40 to 66]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 32 | 44 | 76
  Female | 16 | 40 | 56
  Non-binary | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic | 18 | 38 | 56
  White | 27 | 43 | 70
  Black | 3 | 0 | 3
  Other | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 50 | 86 | 136
Diabetes diagnosis [Count of Participants; unit: Participants] | 14 | 20 | 34
Ureteral stent in place [Count of Participants; unit: Participants] | 13 | 18 | 31
Surgery type [Count of Participants; unit: Participants]
  Ureteroscopy (URS) | 45 | 70 | 115
  Percutaneous | 3 | 14 | 17
  Nephrolithotomy (PCNL) | 2 | 2 | 4
  Other (ESWL or cystolithopaxy) | 0 | 7 | 7
Body Mass Index (BMI) [Median (Full Range); unit: Kg/m^2] | 31 [27 to 35] | 32 [31 to 37] | 32 [27 to 37]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Infection Post Surgery
Description: Number of participants that develop post surgical infection
Time Frame: One to two weeks after surgery (approximately 100 days from baseline)
Population: Patients planning to undergo kidney or bladder stone removal surgery using endoscopy including ureteroscopy and percutaneous nephrolithotomy
Measure: Number; unit: participants
Arm/Group | Intervention Group (NGS + Antibiotic Recommendation) | Control Group
Number analyzed (Participants) | 50 | 86
participants | 0 | 7

2. Secondary Outcome: Number of Participants for Whom Additional Antibiotics Were Selected
Description: The number of participants who required their antibiotic treatment to be augmented (additional antibiotic given) or escalated (broader-spectrum antibiotic chosen).
Time Frame: Within 30 days of urine culture and date of surgery (approximately 100 days from baseline)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group (NGS + Antibiotic Recommendation) | Control Group
Number analyzed (Participants) | 50 | 86
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are collected from Baseline (day 1) up to 90 days from enrollment
Arm/Group | Intervention Group (NGS + Antibiotic Recommendation) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/86
Other Adverse Events (participants affected / at risk) | 0/50 | 1/86
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (NGS + Antibiotic Recommendation) (N=50) | Control Group (N=86)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Hypoglycemia was attributed to a 3 gram dose of cefazolin, the subject presented with a yeast infection.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/55/NCT04404855/Prot_SAP_000.pdf